CLINICAL TRIAL: NCT01880294
Title: CONSIST- Constipation Symptoms Observational Study: A Multicenter, Cross-Sectional Study to Assess Different Diagnostic Criteria of Chronic Constipation in Asia
Brief Title: A Study to Assess Different Diagnostic Criteria of Chronic Constipation in Asia
Acronym: CONSIST
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100891; PRUCOP4003 (Other: Johnson & Johnson Pte Ltd)
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Constipation
Keywords: Constipation; Chronic constipation; Asia-Pacific; Gastroentrology; Asian participants
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Asian participants with chronic constipation: Asian participants diagnosed with chronic constipation using Asian Neurogastro-enterology and Motility Association (ANMA) diagnostic questionnaire.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — Asian participants diagnosed with chronic constipation using ANMA diagnostic questionnaire will be observed.

SUMMARY:
The purpose of the study is to evaluate the differences or similarities in the results obtained with two different scoring systems for chronic constipation in Asian participants consulting in gastroenterology clinics (the Asian Neurogastro-enterology and Motility Association (ANMA) chronic constipation (CC) diagnostic tool (diagnosis questionnaire) and the ROME III diagnosis criteria (western gold standard).

DETAILED DESCRIPTION:
This is an observational (investigators observe participants and measure outcomes without assigning a treatment), non-product specific, regional multicenter (conducted at multiple sites) and multicountry, cross-sectional (observation of all members of a population at one specific point in time), epidemiological study (study of the patterns, causes, and effects of health and disease conditions in defined populations). The study will be conducted in 3 steps. In Step 1 (screening phase), all adult participants visiting their gastroenterologist (for any condition) within a 3 month period will be screened using the ANMA screening worksheet. In Step 2A (diagnosis phase - during investigator chosen consecutive consultation days), all the eligible participants will be required to complete a combination Diagnosis Questionnaire to obtain a diagnosis of CC based on different criteria: self-defined, investigator-judgement, ANMA tool, and ROME III criteria. Details about previous examinations and demography will also be collected during Step 2A of the study, together with Patient Assessment of Constipation Symptoms (PAC-SYM). Participants with a positive response to the ANMA diagnosis tool will proceed to Step 2B. In Step 2B (documentation phase), more information about the participant will be collected using the documentation questionnaire: demography, medical history, history of CC, current symptoms of CC, comorbidities, past and current medications for CC. The Patient Assessment of Constipation-Quality of Life (PAC-QOL) scale will be used to assess participant's satisfaction with their current treatment. Approximately 2000 participants will be screened to yield approximately 400 participants with suspected chronic constipation for whom the Diagnostic and Documentation Questionnaire will be filled in. Safety evaluations will include assessment of adverse events and special reporting situations such as pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have at least 1 of the symptoms listed in the Screening Worksheet and the symptom has been present for at least 3 months
* Participants have signed the informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to complete all the questions on the questionnaires

Exclusion Criteria:

* Participants judged by the investigator to suffer from chronic constipation that is drug-induced or with secondary causes eg, endocrine, metabolic or neurological disorders, surgical obstruction, megacolon/megarectum, a diagnosis of pseudo-obstruction and organic disorders of the large bowel
* Pregnant female participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asian participants diagnosed with chronic constipation using the Asian Neurogastro-enterology and Motility Association diagnostic tool.
Sampling Method: Non-Probability Sample
Enrollment: 461 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2013-12-14 (Actual); Study Completion 2013-12-14 (Actual)

PRIMARY OUTCOMES:
The percentage of participants for whom the chronic constipation (CC) diagnosis, according to the Asian Neurogastro-enterology and Motility Association (ANMA) CC diagnostic tool, agrees with the CC diagnosis according to the ROME III diagnosis criteria | Day 1
  ANMA CC diagnostic criteria: hard stools; difficulty to pass stool; sensation of incomplete evacuation; less than 3 bowel movements per week; straining; sensation of anorectal obstruction; manual maneuvers; CC symptoms for the last 3 months with a symptom onset at least 3 months before diagnosis.
  ROME III CC diagnosis criteria (any 2 or more): straining; lumpy or hard stools; sensation of incomplete evacuation; sensation of anorectal obstruction; manual maneuvers; less than 3 bowel movements per week; CC symptoms for the last 3 months with a symptom onset at least 6 months before diagnosis.
The percentage of participants for whom the CC diagnosis, according to the ANMA CC diagnostic tool, disagrees with the CC diagnosis according to the ROME III diagnosis criteria | Day 1

SECONDARY OUTCOMES:
The percentage of participants with a diagnosis of CC according to the ROME III diagnosis criteria | Day 1
  Number of participants with CC diagnosed by ROME III divided by the number of Asian participants screened (at the gastroenterologist clinic).
The percentage of participants with a diagnosis of CC according to the ANMA CC diagnostic tool | Day 1
  Number of participants with CC diagnosed by ANMA divided by the number of Asian participants screened (at the gastroenterologist clinic).
The percentage of participants with a diagnosis of CC according to investigator judgement | Day 1
  Number of participants with CC diagnosed by investigator's judgement divided by the number of Asian participants screened (at the gastroenterologist clinic).
The percentage of participants with participant self-defined CC | Day 1
  Number of participants with self-defined CC divided by the number of Asian participants screened (at the gastroenterologist clinic).
The percentage of ROME-positive participants who need CC therapy | Day 1
  Number of participants with a positive ROME diagnosis who need CC therapy.
The percentage of ROME-negative but ANMA positive participants who need CC therapy | Day 1
  Number of participants with a negative ROME diagnosis but positive ANMA diagnosis who need CC therapy.
Participant assessment of current treatment as measured by the Constipation-Quality of Life (PAC-QOL) questionnaire | Day 1
  The PAC-QOL is a 28-item scale which includes 4 subscales: worries and concerns, physical discomfort, psychosocial discomfort, and satisfaction. Each item is rated on a 5-point Likert scale ranging from 0 (none of the time or not at all) to 4 (all of the time or extremely). Total score ranges from 0 (best) to 112 (worst). Higher score indicates more impact on QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (14):
- China (4):
  - Beijing
  - Guangzhou
  - Nanjing
  - Wuhan
- Malaysia (2):
  - George Town
  - Kuala Lumpur
- Philippines (3):
  - Manila
  - Quezon City
  - San Juan City
- Singapore, Singapore
- South Korea (4):
  - Daegu
  - Iksan
  - Seongnam-si
  - Seoul